CLINICAL TRIAL: NCT06850506
Title: Exploring the Expression Level of Cadherin 6 Protein (CDH6) in Primary Malignant Bone Tumor Specimens and Its Clinical Application in Prognosis Assessment
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xie Lu, associate chief physician, associate professor, Peking University People's Hospital
Other Study IDs: PKUPH-sarcoma 19
Record Dates: First submitted 2025-01-10; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-12

CONDITIONS: Sarcoma; Sarcoma, Bone; Ewing Sarcoma; Osteosarcoma
Keywords: sarcoma; CDH6; Immunohistochemistry; prognosis; Biological markers
MeSH Terms: conditions — Sarcoma; Osteosarcoma; Sarcoma, Ewing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — Sarcomatous tissue used for immunohistochemistry
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- prechemotherapy: Puncture biopsy or surgical specimens of newly diagnosed patients before chemotherapy
- post-chemotherapy: Conventional chemotherapy regimen

SUMMARY:
1. Evaluate the feasibility of using immunohistochemistry to detect the expression level of CDH6 in histological white slides of patients with osteosarcoma and Ewing's sarcoma as a biological marker for prognostic monitoring The patient's initial visit was clinically diagnosed as high-grade osteosarcoma or Ewing's sarcoma. The informed consent form for specimen monitoring was signed first. During the puncture biopsy, fresh tissue (soft tissue component, not bone tissue) with a volume of about 1cm3 was taken, fixed with formalin solution, and tissue slices (white slices) with a thickness of 5 microns were cut, smeared, and baked. Immunohistochemistry staining was used for CDH6 expression analysis (XP) ® Cadherin-6 (D3T3I) Rabbit mAb Cat:#48111, CellSignaling Technology）。
2. Treatment process and follow-up The routine neoadjuvant chemotherapy regimen for osteosarcoma in our center includes sequential use of cisplatin, high-dose doxorubicin, methotrexate, and ifosfamide, while the VDC-IE regimen is used for Ewing sarcoma (see Figure 3.1.1A, B for details). Due to the significant heterogeneity of osteosarcoma cells, the subpopulations of cells affected by each drug are not the same, and there are also differences in the subpopulations of necrotic and lysed cells after medication. The expression level of CDH6 in patient tissue slices will dynamically change with the sensitivity of chemotherapy. While conducting clinical evaluations, if given the opportunity, we will try to compare the changes in CDH6 levels in tissue sections to assess their value for efficacy monitoring.

   Patients usually undergo surgical treatment after neoadjuvant chemotherapy, and the tumor burden decreases sharply after surgery. The gross tumor specimen obtained during surgery should be retained with qualified tumor tissue samples (at least 1cm3 in volume). During the tumor treatment process, if there is an opportunity for surgery, biopsy or resection of tumor tissue should be performed again to monitor changes in CDH6 expression levels. Clinical evaluation of tumor treatment should be conducted every two months until the end of the study or patient death.

   The entire study includes a screening period, blood collection and specimen retention period, and follow-up period. All participants in the study must meet all inclusion and exclusion criteria.

   During the screening period, potential participants will undergo eligibility assessment for the study after signing the informed consent form. Subjects must undergo radiographic evaluation of the disease within 14 days prior to neoadjuvant chemotherapy, including enhanced CT or MRI of the primary tumor site, chest plain scan CT, ECT whole-body bone imaging, or whole-body PET/CT.

   The subjects will receive chemotherapy and surgical treatment according to the diagnosis and treatment routine, and at the time nodes designed in the experiment, before and after the subjects' routine chemotherapy and surgery, the pathology department will take 3 white slides, each measuring 4 microns, smear and bake gel, and perform immunohistochemical staining.

   During the follow-up period, the subjects have completed chemotherapy and surgical treatment, but will still receive follow-up on their survival status and oncology status, and all follow-up will be routine treatment at our center.
3. We will use FFPE tumor tissue samples for immunohistochemical staining to analyze the expression of CDH6, β - catenin, and CDH17 in tumor tissue.

Immunohistochemical staining:

Primary antibody: CDH6 rabbit monoclonal antibody (D3T3I); β - catenin rabbit monoclonal antibody (D10A8); CDH17 mouse monoclonal antibody (Xianxiang internal antibody); Secondary antibody detection system: Bond Polymer Refine Detection Kit； Antibody diluent: CST,8112L,#38； Positive photos: FFPE sections of low, medium, and high expression cell lines; The staining program uses the established method of Xianxiang.

Pathological interpretation:

Use H-score for semi quantitative analysis. H-score is the sum of the percentage of cell staining multiplied by the corresponding intensity values (0=negative, 1=1+, 2=2+, 3=3+), ranging from 0 to 300.

The interpretation of tumor cell staining intensity values is as follows:

High expression (3+): Strong cell membrane staining and/or cytoplasmic staining were observed under x4 magnification; Moderate expression (2+): Cell membrane staining was observed at x10 or x20 magnification; Low expression (1+): weak cell membrane staining and/or cytoplasmic staining were observed at x40 magnification; Negative (0): No cell membrane staining and/or cytoplasmic staining was observed in tumor cells.

DETAILED DESCRIPTION:
1. Evaluate the feasibility of using immunohistochemistry to detect the expression level of CDH6 in histological white slides of patients with osteosarcoma and Ewing's sarcoma as a biological marker for prognostic monitoring The patient's initial visit was clinically diagnosed as high-grade osteosarcoma or Ewing's sarcoma. The informed consent form for specimen monitoring was signed first. During the puncture biopsy, fresh tissue (soft tissue component, not bone tissue) with a volume of about 1cm3 was taken, fixed with formalin solution, and tissue slices (white slices) with a thickness of 5 microns were cut, smeared, and baked. Immunohistochemistry staining was used for CDH6 expression analysis (XP) ® Cadherin-6 (D3T3I) Rabbit mAb Cat:#48111, CellSignaling Technology）。
2. Treatment process and follow-up The routine neoadjuvant chemotherapy regimen for osteosarcoma in our center includes sequential use of cisplatin, high-dose doxorubicin, methotrexate, and ifosfamide, while the VDC-IE regimen is used for Ewing sarcoma (see Figure 3.1.1A, B for details). Due to the significant heterogeneity of osteosarcoma cells, the subpopulations of cells affected by each drug are not the same, and there are also differences in the subpopulations of necrotic and lysed cells after medication. The expression level of CDH6 in patient tissue slices will dynamically change with the sensitivity of chemotherapy. While conducting clinical evaluations, if given the opportunity, we will try to compare the changes in CDH6 levels in tissue sections to assess their value for efficacy monitoring.

   Patients usually undergo surgical treatment after neoadjuvant chemotherapy, and the tumor burden decreases sharply after surgery. The gross tumor specimen obtained during surgery should be retained with qualified tumor tissue samples (at least 1cm3 in volume). During the tumor treatment process, if there is an opportunity for surgery, biopsy or resection of tumor tissue should be performed again to monitor changes in CDH6 expression levels. Clinical evaluation of tumor treatment should be conducted every two months until the end of the study or patient death.

   The entire study includes a screening period, blood collection and specimen retention period, and follow-up period. All participants in the study must meet all inclusion and exclusion criteria.

   During the screening period, potential participants will undergo eligibility assessment for the study after signing the informed consent form. Subjects must undergo radiographic evaluation of the disease within 14 days prior to neoadjuvant chemotherapy, including enhanced CT or MRI of the primary tumor site, chest plain scan CT, ECT whole-body bone imaging, or whole-body PET/CT.

   The subjects will receive chemotherapy and surgical treatment according to the diagnosis and treatment routine, and at the time nodes designed in the experiment, before and after the subjects' routine chemotherapy and surgery, the pathology department will take 3 white slides, each measuring 4 microns, smear and bake gel, and perform immunohistochemical staining.

   During the follow-up period, the subjects have completed chemotherapy and surgical treatment, but will still receive follow-up on their survival status and oncology status, and all follow-up will be routine treatment at our center.
3. We will use FFPE tumor tissue samples for immunohistochemical staining to analyze the expression of CDH6, β - catenin, and CDH17 in tumor tissue.

Immunohistochemical staining:

Primary antibody: CDH6 rabbit monoclonal antibody (D3T3I); β - catenin rabbit monoclonal antibody (D10A8); CDH17 mouse monoclonal antibody (Xianxiang internal antibody); Secondary antibody detection system: Bond Polymer Refine Detection Kit； Antibody diluent: CST,8112L,#38； Positive photos: FFPE sections of low, medium, and high expression cell lines; The staining program uses the established method of Xianxiang.

Pathological interpretation:

Use H-score for semi quantitative analysis. H-score is the sum of the percentage of cell staining multiplied by the corresponding intensity values (0=negative, 1=1+, 2=2+, 3=3+), ranging from 0 to 300.

The interpretation of tumor cell staining intensity values is as follows:

High expression (3+): Strong cell membrane staining and/or cytoplasmic staining were observed under x4 magnification; Moderate expression (2+): Cell membrane staining was observed at x10 or x20 magnification; Low expression (1+): weak cell membrane staining and/or cytoplasmic staining were observed at x40 magnification; Negative (0): No cell membrane staining and/or cytoplasmic staining was observed in tumor cells.

ELIGIBILITY:
Inclusion Criteria:

1. Over 12 years old.
2. High grade osteosarcoma or Ewing's sarcoma confirmed by clinical judgment or histopathology. Patients with local tumors and isolated lesions in the lungs must obtain pathological diagnosis confirmation, while multiple metastases in the lungs do not require pathological examination.
3. Newly diagnosed patients who have not received formal first-line chemotherapy for osteosarcoma or Ewing's sarcoma. (First line chemotherapy drugs include high-dose methotrexate, anthracyclines, cisplatin, and ifosfamide; the first-line treatment regimen for Ewing's sarcoma is VDC sequential IE.)
4. All other examination indicators suggest that standardized chemotherapy and surgical treatment for bone tumors can be accepted.

Exclusion Criteria:

1. Cannot accept standardized chemotherapy and surgical treatment for bone tumors in our center.
2. Not accepting standardized diagnosis and treatment routine follow-up.
3. The researcher believes that there are any conditions that may harm the subjects or cause them to be unable to meet or perform the research requirements.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 70 patients with osteosarcoma or Ewing's sarcoma
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
CDH6 protein expression | Baseline
  Immunochemotherapy

SECONDARY OUTCOMES:
tumor necrosis rate | Within 24 hours after surgery
  Pathological microscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No